CLINICAL TRIAL: NCT05157932
Title: An Evaluation of the Talk Test as an Effective and Safe Approach for Exercise Prescription for Home-Based Cardiac Rehabilitation: A Pilot RCT
Brief Title: An Evaluation of the Talk Test for Exercise Prescription for Home-Based Cardiac Rehabilitation
Acronym: Talk-Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20210525-01H
Record Dates: First submitted 2021-10-08; First posted 2021-12-15 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Talk test; Cardiopulmonary Exercise test; Cardiac rehabilitation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Talk Test (Experimental): Virtual Cardiac Rehab + Exercise prescription based on the Talk test.
  Interventions: Behavioral: Talk test prescription
- Cardiopulmonary Exercise Test (Experimental): Virtual Cardiac Rehab + Exercise prescription based on the CPET results.
  Interventions: Behavioral: CPET prescription

INTERVENTIONS:
Behavioral: Talk test prescription — Participants will be enrolled in the virtual cardiac rehab program and receive an exercise prescription based on the Talk test method.
  Arms: Talk Test
Behavioral: CPET prescription — Participants will be enrolled in the virtual cardiac rehab program and receive an exercise prescription based on their CPET results completed at baseline
  Arms: Cardiopulmonary Exercise Test

SUMMARY:
The objectives of this pilot RCT are to examine if the Talk Test is an effective and safe tool as compared with CPET for exercise prescription in patients who have undergone CABG or PCI and enrolled in a home-based CR program with virtual exercise training monitoring.

DETAILED DESCRIPTION:
The Talk Test has been shown to be a valid, practical and inexpensive tool for guiding exercise training in patients with CAD. The general premise of the Talk Test is that exercising at or above the ventilatory threshold or lactate threshold does not allow comfortable, conversational speech and thus serves as a means of estimating the cut point between moderate and vigorous intensity exercise. The Talk Test can be used to produce exercise intensities (64 to 95% HR peak i.e. moderate-to-vigorous intensity exercise) within accepted Canadian Association of Cardiovascular Prevention and Rehabilitation (CACPR) guidelines for exercise training, to avoid exertional ischemia, and has been shown to be consistent across various modes of exercise (i.e. walking, jogging, cycling, elliptical trainer and stair stepper).

There is a critical need to evaluate the effectiveness and safety of using the Talk Test as the principal method of exercise prescription in patients with CAD who have undergone CABG or PCI when compared to standard care CPET. Such a trial has wide-scale appeal for CR programs across Canada and beyond. It will directly and positively impact patient care by reducing the need for in-person interactions for CPET, of paramount importance during COVID-19 outbreaks, between patients and CR staff, thus reducing COVID-19 infection risk and concerns of contracting the virus.

ELIGIBILITY:
Inclusion Criteria:

* recently underwent PCI or CABG (at least 4 weeks but less than 12 weeks post-event or procedure);
* able to perform a CPET;
* at least 40 years of age;
* access to MyChart; and,
* access to email and the internet
* access to a cellphone with broadband internet (4G, LTE, 5G).

Exclusion Criteria:

* currently participating in a virtual or on-site CR program;
* ventricular ejection fraction ≤45%;
* unstable angina or established diagnosis of chronic obstructive pulmonary disease, severe mitral or aortic stenosis, or hypertrophic obstructive cardiomyopathy;
* unable to return for 12-week follow-up visits.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | from baseline to follow-up at week 12
  will be measured by the Incremental Shuttle Walk Test.

SECONDARY OUTCOMES:
Cardiovascular health indicators - Plasma glucose | from baseline to follow-up at week 12
  will be measured by fasting plasma glucose (mmol/L) test
Cardiovascular health indicators - Plasma glucose average | from baseline to follow-up at week 12
  will be measured using the glycated hemoglobin A1C (%) test
Cardiovascular health indicators - Lipid profile | from baseline to follow-up at week 12
  will be measured using the triglycerides test
Cardiovascular health indicators - Cholesterol HDL | from baseline to follow-up at week 12
  will be measured high-density lipoprotein cholesterol.
Cardiovascular health indicators - Cholesterol LDL | from baseline to follow-up at week 12
  will be measured low-density lipoprotein cholesterol.
Cardiac Rehab safety | from baseline to follow-up at week 12
  meticulously track all mild, moderate, and severe symptoms and adverse events throughout this study. Symptoms may include tightness in chest, leg tightness/pain, dizziness, lightheaded, foot cramping, and heart palpitations.
VO2peak | at baseline
  will be measured using a gold standard symptom-limited CPET on an electronically braked cycle ergometer (alternatively it will be administered on a treadmill or another aerobic equipment). Gas exchange (VO2 in mL/kg/min) and heart rate will be monitored continuously. The highest 20-s interval average of VO2 and HR will be considered the peak VO2 and HR values.

OTHER OUTCOMES:
Exercise prescription compliance | from baseline to follow-up at week 12
  Talk Test group: HR will be measured during exercise training using the Polar A370 device. Following each exercise session, participants will record on a Talk Test log if: (1) singing was possible, (2) comfortable conversation, but not singing was possible, or (3) comfortable conversation was not possible. These responses will be coded as "does not comply", "complies" and "exceeds". CPET group: HR will be measured during exercise training using the Polar A370 device. Where participants exercise below, within or above the prescribed HR ranges (64 to 95% HR peak), they will be coded as "does not comply", "complies" and "exceeds". All participants will wear Polar A370 devices during their exercise training sessions. Exercise HRs will be compared between the Talk Test and CPET groups.
Cardiometabolic health indicators - BMI | from baseline to follow-up at week 12
  Height (cm) and body mass (kg) will be measured to compute body mass index (kg/m2)
Cardiometabolic health indicators - Body composition | from baseline to follow-up at week 12
  Body composition will be measured using Fat mass (%) and fat-free mass (%), using bioelectrical impedance analysis.
Cardiometabolic health indicators - Cardiometabolic Risk | from baseline to follow-up at week 12
  will be measured using waist circumference (cm) and will be measured using standardized procedures.
Cardiometabolic health indicators - Blood pressure | from baseline to follow-up at week 12
  Resting Systolic (mmHg) and Diastolic (mmHg) blood pressure will be measured in a seated position after a 5-minute rest period on the right arm using an automated, BP monitor (BPTru) that measures 6 times (the first will be discarded and an average of the last 5 measurements will be used for statistical analyses) at 2-minute intervals.
Gender | from baseline to follow-up at week 12
  gender and its effect will be assessed during cardiac rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pipe, MD, Study Chair — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
it is not yet known if there will be a plan to make IPD available.